CLINICAL TRIAL: NCT05127343
Title: One Year Clinical Comparison Between Resin Based and Glass Ionomer Based Hydrophilic Fissure Sealants Among Adolescents: A Randomized Clinical Trial
Brief Title: Comparison Between Resin Based and Glass Ionomer Based Hydrophilic Fissure Sealants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Mohamed El-Amir Hashim Sediek, Master's Degree student- Faculty of Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CU-2021
Record Dates: First submitted 2021-11-12; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Caries
Keywords: Pit and fissure sealant; Retention rate; Caries formation; Hydrophilic sealant
MeSH Terms: conditions — Van der Woude syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resin based sealant (Ultraseal XT Hydro) (Active Comparator)
  Interventions: Procedure: Sealing deep pits and fissures
- Glass ionomer based sealant (Fugi Triage) (Active Comparator)
  Interventions: Procedure: Sealing deep pits and fissures

INTERVENTIONS:
Procedure: Sealing deep pits and fissures — Application of the pit and fissure sealant

SUMMARY:
The aim of the study is to clinically evaluate the retention and caries formation of hydrophilic fissure sealants among adolescents after one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have existing pits and fissures that are anatomically deep and caries susceptible.
* Healthy patients with no history of previous systematic diseases that can affect their oral health and sealant application.
* Cooperative patients who will allow the clinical applications

Exclusion Criteria:

* Uncooperative behaviour limiting the use of sealants throughout the procedure.
* Patients with history of medical diseases, drug therapies or any other serious relevant problem.
* Patients with well coalesced pits and fissures
* Patients allergic to sealant material
* Patients who underwent orthodontic treatment.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Retention rate | Change from baseline at 3, 6, 12 months
  * Full retention (FR): The material is fully present on the occlusal surfaces
  * Partially lost (PL): The material is present, but as a result of either wear or loss of the material, part of the previously sealed fissure, was exposed.
  * Totally lost (TL): No trace of the material to be detected on the surface

SECONDARY OUTCOMES:
Caries formation | Change from baseline at 3, 6, 12 months
  Decayed: If the explorer caught on the tooth after insertion into the fissures

CONTACTS AND LOCATIONS:
Overall Officials: Iman I ElSayad, Professor, Study Director — Cairo University; Heba Helal, Study Director — Cairo University
Locations (1):
- Faculty of dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided